CLINICAL TRIAL: NCT02792075
Title: Prognosis of Coronary Stenosis Based on Intracoronary Imaging; A Multicenter, Prospective Observational Study
Acronym: IRIS imaging
Status: Recruiting | Type: Observational
Sponsor: Seung-Jung Park (Other)
Collaborators: CardioVascular Research Foundation, Korea (Other)
Responsible Party: Sponsor-Investigator, Seung-Jung Park, professor of medicine, Asan Medical Center
Organization: Asan Medical Center (Other)
Other Study IDs: AMCCV2016-09
Record Dates: First submitted 2016-06-02; First posted 2016-06-07 (Estimated); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Coronary Artery Disease
Keywords: Coronary Stenosis; Intracoronary Imaging; VH-IVUS; OCT; NIRS; gray scale IVUS
MeSH Terms: conditions — Coronary Artery Disease; Coronary Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- VH-IVUS: Patients with IVUS-derived virtual histology
  Interventions: Other: 5-year Follow-up
- OCT: Patients with Optical coherence tomography
  Interventions: Other: 5-year Follow-up
- NIRS: Patients with Near-infrared spectroscopy
  Interventions: Other: 5-year Follow-up
- gray scale IVUS: Patients with gray-scale IVUS(Intravascular ultrasound)
  Interventions: Other: 5-year Follow-up

INTERVENTIONS:
Other: 5-year Follow-up

SUMMARY:
The purpose of this study is to evaluate the prognosis of coronary stenosis based on intracoronary Imaging.

ELIGIBILITY:
Inclusion Criteria:

* Patients with intracoronary imaging
* Written consent

Exclusion Criteria:

* Severe calcification and/or severe tortuosity
* Lesion with previous bypass graft surgery (CABG)
* Left ventricular ejection fraction less than 30 %
* Coronary spasm
* Life expectancy less than 2 years
* Pregnancy or breast-feeding

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with intracoronary imaging
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2016-07 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2030-06 (Estimated)

PRIMARY OUTCOMES:
Target Vessel Failure | 2 years
  defined as composite event of cardiac death, non-fatal myocardiac infarction, target vessel revascularization

SECONDARY OUTCOMES:
All-cause death | 5 years
Cardiac death | 5 years
Number of myocardial infarction events | 5 years
  Q wave myocardial infarction or non Q wave myocardial infarction
Composite event of death or myocardial infarction | 5 years
Composite event of cardiac death or myocardial infarction | 5 years
Target Vessel revascularization | 5 years
Target Lesion revascularization | 5 years
Number of stent thrombosis events | 5 years
  DEFINITE stent thrombosis : acute coronary syndrome and angiographic or pathologic evidence of stent thrombosis; PROBABLE stent thrombosis : unexplained death within 30 days or target-vessel infarction without angiographic information Academic Research Consortium (ARC) stent thrombosis is reported as a cumulative value at different time points and within the different separate time points. Time 0 is the time point after the guide catheter has been removed. Acute stent thrombosis: 0-24 hours after stent implantation; Subacute stent thrombosis: >24 hours to 30 days post; late stent thrombosis: >30 days to 1 year post; Very late stent thrombosis: >1 year post;
Number of stroke | 5 years
Procedural success | 7 days
  Defined as mean lesion diameter stenosis less than 30% and without the occurrence of in-hospital myocardial infarction (MI), target vessel revascularization (TVR), or death

CONTACTS AND LOCATIONS:
Locations (15):
- South Korea (15):
  - Asan Medical Center, Seoul, Songpa-gu
  - Inje University Busan Paik Hospital, Busan
  - Soon Chun Hyang University Hospital Cheonan, Cheonan
  - Keimyung University Dongsan Medical Center, Daegu
  - Chungnam National University Hospital, Daejeon
  - Inje University Ilsan Paik Hospital, Ilsan
  - Gachon University Gil Hospital, Incheon
  - Jeju national university hospital, Jeju City
  - Pusan National University Hospital, Pusan
  - Chung-Ang university hospital, Seoul
  - Kangbuk Samsung Hospital, Seoul
  - Korea University Guro Hospital, Seoul
  - Ajou University Hospital, Suwon
  - Ulsan University Hospital, Ulsan
  - Wonju Severance Christian Hospital, Wŏnju

IPD SHARING:
Plan to Share IPD: No
This is not a publicly funded trial.